CLINICAL TRIAL: NCT06800703
Title: Opioid Use Disorder and Pain
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Brain and Behavior Research Foundation (previously known as NARSAD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2000039121; 4R00AA029716-03 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-30 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder; Healthy Controls Group - Age and Sex-matched
Keywords: opioid use disorder; pain; avoidance learning; prediction
MeSH Terms: conditions — Opioid-Related Disorders; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- opioid use disorder: individuals with OUD diagnosis
  Interventions: Behavioral: follow up interviews for 12 months to determine opioid use
- Healthy controls: Healthy individuals without substance use disorders

INTERVENTIONS:
Behavioral: follow up interviews for 12 months to determine opioid use — Follow-up
  Groups: opioid use disorder

SUMMARY:
The goal of this observational study is to characterize the brain processes of pain avoidance learning dysfunctions in individuals with opioid use disorder (OUD). The main questions it aims to answer are:

Compared with healthy controls, do those with OUD exhibit impaired avoidance learning in response to pain? What are the brain processes that are associated with this avoidance learning dysfunction? Do these brain processes serve to predict future use or relapse?

Researchers will compare those with OUD and healthy controls to determine avoidance learning dysfunction and its relationship with opioid use.

Participants will be performing a learning task inside an fMRI scanner. Those with OUD will also be followed up for a year to determine future opioid use.

DETAILED DESCRIPTION:
Opioid Use Disorder (OUD) is a chronic condition with exceptionally high relapse rates. Over 80% of patients receiving treatment relapse within a year. To understand the etiological processes of OUD, investigators have focused on reward seeking as a primary drinking motive. However, whereas reward and sensation seeking may be central to the early stages of OUD, it is posited that drinking as an avoidance coping behavior plays a more critical role in the maintenance of OUD. Specifically, as opioid escalates, consumption is increasingly driven by individuals' enhanced sensitivity to the aversive consequences of withdrawal. This indicates a fundamental shift of motivation from positive to negative reinforcement in OUD. Paradoxically, while users seek opioid to avoid painful physical and emotional states, chronic opioid use heightens pain reactivity, which further motivates drug use as an avoidance coping strategy. Over time, this maladaptive behavior becomes progressively less amenable to cognitive control, trapping users in a spiraling cycle of drug use and distress. The investigators thus hypothesize that dysfunctional avoidance learning is a central pathophysiological process of OUD.

Avoidance learning is a product of pain reactivity and cognitive control and their underlying brain circuits. Yet, how avoidance learning and its circuit processes are compromised in individuals with OUD remains unclear. This study aims to fill this important gap in research by investigating avoidance learning deficits as a principal mechanism of OUD.

The current proposal leverages neuroimaging, physiological recordings, and clinical assessments of avoidance learning to identify a set of markers to distinguish those with OUD from healthy controls (HC), evaluate the "diagnostic" accuracy of these markers, and describe how they may predict relapse. The investigators will also examine reward learning as a contrast to differentiate its role in OUD. Avoidance and reward learning will be operationalized via a probabilistic learning go/no-go task in which participants learn to associate cues with outcomes to avoid electric shocks and optimize reward. First, the investigators will identify brain dysfunctions in avoidance and reward learning in OUD patients and establish their inter-relationships with clinical and drug use characteristics. Next, in addition to continuing recruitment, the investigators will follow up with OUD patients for 12 months to identify predictors of relapse. The investigators will also follow up with opioid regular users to determine changes in opioid use over time.

Individuals with OUD and HCs will be recruited from the Greater New Haven, Hartford, Bridgeport areas of CT. Those with OUD will be drawn by self-referral based on seeing flyers and brochures posted at treatment programs such as the Substance Abuse Treatment Unit (SATU) and the Connecticut Mental Health Center (CMHC), by advertisements of the study, or by word of mouth. HCs will be recruited from the community by flyers and advertisements or by word of mouth.

Ninety treatment-seeking individuals with OUD (45 women) between 21 and 60 years of age and meeting the diagnosis of moderate to severe OUD will be recruited to participate in the study.

Forty individuals with regular opioid use (i.e., at least weekly, non-prescription) (20 women) aged between 21-60 who are not seeking treatment will also be recruited.

Ninety HCs (45 women) with matching demographics (including age, sex, race, and education) will be recruited. HCs will undergo the same intake assessments to confirm eligibility.

ELIGIBILITY:
Patients with Opioid Use Disorder (OUD)

To be eligible for inclusion in the study, an individual must meet all of the following criteria:

1. Between ages 21-60 years old.
2. Able to read and write and provide written informed consent.
3. Meet DSM-5 criteria for moderate to severe opioid use disorder; self-reported excessive opioid use prior to study entry and verified by urine toxicology testing; seeking treatment for their OUD.
4. Physically healthy with no major medical illnesses, history of head injury or any neurological illness
5. No plans to relocate out of state in the next 12 months (for follow-up purposes).
6. Currently seeking treatment or currently receiving treatment for OUD.
7. Speak English
8. Have been enrolled in an inpatient or outpatient treatment program for OUD for at least 4 weeks.

Exclusion Criteria:

1. Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, hepatic, thyroid pathology.
2. History of head injury with loss of consciousness (> 30 minutes).
3. Current or past DSM-IV or DSM 5 diagnosis of a major psychiatric disorder (other than opioid and nicotine use disorders) that required hospitalization, or that required daily medications for over 4 weeks. Such medications include antidepressants, anticholinergics, antipsychotics, anxiolytics, lithium, psychotropic drugs not otherwise specified including herbal products, drugs with psychomotor effects or with anxiolytics, stimulant, or antipsychotic properties, any other psychoactive drugs, and sedatives/hypnotics. Individuals with current depressive or anxiety symptoms requiring treatment or currently being treated for these symptoms will be excluded.
4. Any subjects with foreign ferromagnetic metal objects in their body or other MR contraindications will be excluded. Individuals who previously worked in metal industry or with metal shavings (due to a risk of any remaining metal particles moving in the eye during the MRI).
5. Pregnant or lactating women will not be recruited for the study.
6. Cannot or are not willing to lie comfortably flat on his/her back for up to 2 hours in the MRI scanner (self-report).
7. Body weight > 550 lbs. The MR scanner bed is tested to a weight limit of 550 lbs.
8. No pPlans to relocate out of state in the next 12 months (for follow-up purposes).
9. Still experiencing significant withdrawal symptoms.

Individuals with regular opioid use

To be eligible for inclusion in the study, an individual must meet all of the following criteria:

1. Between ages 21-60 years old.
2. Able to read and write and provide written informed consent.
3. Use non-prescribed opioids on a weekly basis or more.
4. Physically healthy with no major medical illnesses, history of head injury or any neurological illness
5. No plans to relocate out of state in the next 12 months (for follow-up purposes).
6. Speak English

Exclusion Criteria:

1. Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, hepatic, thyroid pathology.
2. History of head injury with loss of consciousness (> 30 minutes).
3. Current or past DSM-IV or DSM 5 diagnosis of a major psychiatric disorder (other than opioid and nicotine use disorders) that required hospitalization, or that required daily medications for over 4 weeks. Such medications include antidepressants, anticholinergics, antipsychotics, anxiolytics, lithium, psychotropic drugs not otherwise specified including herbal products, drugs with psychomotor effects or with anxiolytics, stimulant, or antipsychotic properties, any other psychoactive drugs, and sedatives/hypnotics. Individuals with current depressive or anxiety symptoms requiring treatment or currently being treated for these symptoms will be excluded.
4. Any subjects with foreign ferromagnetic metal objects in their body or other MR contraindications will be excluded.
5. Pregnant or lactating women will not be recruited for the study.
6. Cannot or are not willing to lie comfortably flat on his/her back for up to 2 hours in the MRI scanner (self-report).
7. Body weight > 550 lbs. The MR scanner bed is tested to a weight limit of 550 lbs.

Individuals with regular opioid use

To be eligible for inclusion in the study, an individual must meet all of the following criteria:

1. Between ages 21-60 years old.
2. Able to read and write and provide written informed consent.
3. Use non-prescribed opioids on a weekly basis or more.
4. Physically healthy with no major medical illnesses, history of head injury or any neurological illness
5. No plans to relocate out of state in the next 12 months (for follow-up purposes).
6. Speak English

Exclusion Criteria:

1. Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, hepatic, thyroid pathology.
2. History of head injury with loss of consciousness (> 30 minutes).
3. Current or past DSM-IV or DSM 5 diagnosis of a major psychiatric disorder (other than opioid and nicotine use disorders) that required hospitalization, or that required daily medications for over 4 weeks. Such medications include antidepressants, anticholinergics, antipsychotics, anxiolytics, lithium, psychotropic drugs not otherwise specified including herbal products, drugs with psychomotor effects or with anxiolytics, stimulant, or antipsychotic properties, any other psychoactive drugs, and sedatives/hypnotics. Individuals with current depressive or anxiety symptoms requiring treatment or currently being treated for these symptoms will be excluded.
4. Any subjects with foreign ferromagnetic metal objects in their body or other MR contraindications will be excluded.
5. Pregnant or lactating women will not be recruited for the study.
6. Cannot or are not willing to lie comfortably flat on his/her back for up to 2 hours in the MRI scanner (self-report).
7. Body weight > 550 lbs. The MR scanner bed is tested to a weight limit of 550 lbs.

Individuals with regular opioid use

To be eligible for inclusion in the study, an individual must meet all of the following criteria:

1. Between ages 21-60 years old.
2. Able to read and write and provide written informed consent.
3. Use non-prescribed opioids on a weekly basis or more.
4. Physically healthy with no major medical illnesses, history of head injury or any neurological illness
5. No plans to relocate out of state in the next 12 months (for follow-up purposes).
6. Speak English

Exclusion Criteria:

1. Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, hepatic, thyroid pathology.
2. History of head injury with loss of consciousness (> 30 minutes).
3. Current or past DSM-IV or DSM 5 diagnosis of a major psychiatric disorder (other than opioid and nicotine use disorders) that required hospitalization, or that required daily medications for over 4 weeks. Such medications include antidepressants, anticholinergics, antipsychotics, anxiolytics, lithium, psychotropic drugs not otherwise specified including herbal products, drugs with psychomotor effects or with anxiolytics, stimulant, or antipsychotic properties, any other psychoactive drugs, and sedatives/hypnotics. Individuals with current depressive or anxiety symptoms requiring treatment or currently being treated for these symptoms will be excluded.
4. Any subjects with foreign ferromagnetic metal objects in their body or other MR contraindications will be excluded.
5. Pregnant or lactating women will not be recruited for the study.
6. Cannot or are not willing to lie comfortably flat on his/her back for up to 2 hours in the MRI scanner (self-report).
7. Body weight > 550 lbs. The MR scanner bed is tested to a weight limit of 550 lbs.

Healthy controls (HC) Inclusion Criteria

1. Between ages 1821-60 years old.
2. Able to read and write and provide written informed consent.
3. Demographics matching OUD participants.
4. Speak English

Exclusion Criteria:

1. Meet criteria for current or history of any Axis I (except nicotine use) disorder.
2. Any significant current medical condition such as neurological, cardiovascular, endocrine, renal, hepatic, thyroid pathology. History of head injury with loss of consciousness (> 30 minutes).

4. Any subjects with foreign ferromagnetic metal objects in their body or other MR contraindications will be excluded.

5. Pregnant or lactating women will not be recruited for the study. 6. Cannot or are not willing to lie comfortably flat on his/her back for up to 2 hours in the MRI scanner (self-report).

7. Body weight > 550 lbs. The MR scanner bed is tested to a weight limit of 550 lbs.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Treatment-seeking OUD patients will be recruited from local clinics. Those with OUD not seeking treatment and healthy controls will be recruited from New Haven and surrounding areas in Connecticut.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Avoidance learning measure | Day 1 (immediately after consent and clinical assessment)
  Task performance measure of avoidance learning, quantified by response time and performance accuracy. Those with OUD are expected to have lower performance accuracy, lower learning rates, and higher response time during avoidance learning relative to healthy controls
opioid use | During the 12-month follow-up period
  Quantity of opioid use following the baseline visit, measured by times use per week. Timeline follow back method will be used to assess the quantity of opioid use during the follow-up period. The investigators will examine this opioid use quantity in relation with avoidance learning deficits. The investigators expect greater avoidance dysfunction at baseline to predict higher weekly use of opioids
Brain activity during avoidance learning | Day 1 (immediately after consent and clinical assessment)
  The brain activation magnitude associated with avoidance learning and avoidance learning dysfunction during the task performance. Brain activation will be computed by using contrast between avoidance learning vs. neutral conditions. Contrasts between two subject groups (i.e., OUD vs. HC) will also be examined. The investigators expect OUD patients to exhibit greater activations in the pain circuit during avoidance learning relative to healthy controls. Additionally, pain circuit activation will be assessed in association with opioid use severity during follow-up period.

SECONDARY OUTCOMES:
Comparison of avoidance learning rate between women and men | Day 1 (immediately after consent and clinical assessment)
  Sex differences in avoidance learning dysfunction in those with opioid use disorder. Comparison between women and men will be conducted in relation to their avoidance learning task performance (e.g., performance accuracy, response time)
Comparison of brain activity during avoidance learning between women and men | Day 1 (immediately after consent and clinical assessment)
  Comparison between women and men will be conducted in relation to their brain activations during avoidance learning to determine whether women or men may have higher brain activity amplitude during learning of avoidance behavior.
Relationship between sex differences in avoidance learning and opioid use | Day 1 (immediately after consent and clinical assessment)
  Investigators will examine whether opioid use severity has a relationship with differences in avoidance learning performance.

CONTACTS AND LOCATIONS:
Overall Officials: Thang M Le, PhD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, S105, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD at this time

REFERENCES:
- [Result] Baker TB, Piper ME, McCarthy DE, Majeskie MR, Fiore MC. Addiction motivation reformulated: an affective processing model of negative reinforcement. Psychol Rev. 2004 Jan;111(1):33-51. doi: 10.1037/0033-295X.111.1.33. PMID 14756584
- [Result] Carcoba LM, Contreras AE, Cepeda-Benito A, Meagher MW. Negative affect heightens opiate withdrawal-induced hyperalgesia in heroin dependent individuals. J Addict Dis. 2011 Jul-Sep;30(3):258-70. doi: 10.1080/10550887.2011.581985. PMID 21745048
- [Result] Ren ZY, Shi J, Epstein DH, Wang J, Lu L. Abnormal pain response in pain-sensitive opiate addicts after prolonged abstinence predicts increased drug craving. Psychopharmacology (Berl). 2009 Jun;204(3):423-9. doi: 10.1007/s00213-009-1472-0. Epub 2009 Jan 27. PMID 19172249
- [Result] Grella CE, Lovinger K. 30-year trajectories of heroin and other drug use among men and women sampled from methadone treatment in California. Drug Alcohol Depend. 2011 Nov 1;118(2-3):251-8. doi: 10.1016/j.drugalcdep.2011.04.004. Epub 2011 May 6. PMID 21549528
- [Result] Le TM, Zhornitsky S, Wang W, Zhang S, Li CR. Problem drinking alters gray matter volume and food cue responses of the lateral orbitofrontal cortex. Addict Biol. 2021 Jan;26(1):e12857. doi: 10.1111/adb.12857. Epub 2019 Nov 20. PMID 31746092
- [Result] Wang W, Zhornitsky S, Le TM, Zhang S, Li CR. Heart Rate Variability, Cue-Evoked Ventromedial Prefrontal Cortical Response, and Problem Alcohol Use in Adult Drinkers. Biol Psychiatry Cogn Neurosci Neuroimaging. 2020 Jun;5(6):619-628. doi: 10.1016/j.bpsc.2019.12.013. Epub 2019 Dec 30. PMID 32061544
- [Result] Le TM, Chao H, Levy I, Li CR. Age-Related Changes in the Neural Processes of Reward-Directed Action and Inhibition of Action. Front Psychol. 2020 Jun 10;11:1121. doi: 10.3389/fpsyg.2020.01121. eCollection 2020. PMID 32587547
- [Result] Le TM, Zhang S, Zhornitsky S, Wang W, Li CR. Neural correlates of reward-directed action and inhibition of action. Cortex. 2020 Feb;123:42-56. doi: 10.1016/j.cortex.2019.10.007. Epub 2019 Oct 31. PMID 31747630